CLINICAL TRIAL: NCT06267573
Title: Outcomes of Endovascular Repair of Thoracoabdominal Aortic Aneurysms
Brief Title: Thoracoabdominal Aortic Aneurysms
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Raafat Khalil Gad, Assistant lecturer, Assiut University
Other Study IDs: Kerolos protocol
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Fenestrated and branched endovascular devices for TAAA — Devices for TAAA

SUMMARY:
Evaluation of the effectiveness of the different modalities for treatment of thoracoabdominal aortic aneurysms. FEVAR and BEVAR devices are widely used now due to its feasability and wide range of use . We aim to evaluate the effectiveness of these new devices in the management of TAAA

ELIGIBILITY:
Inclusion Criteria:

* all adult consecutive patients presenting with TAAA larger than 5.5 cm

Exclusion Criteria:

* active infection Asymptomatic patients with small aneurysms Allergy to contrast agents

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Successful cannulation of the target vessels with complete in-line flow to target organs. | Two years
  No ischemia

IPD SHARING:
Plan to Share IPD: No